CLINICAL TRIAL: NCT01952977
Title: Effect of Medium Chain Triglyceride Consumption on Appetite
Acronym: MCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Research Associate, St. Luke's-Roosevelt Hospital Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MCT_1
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCT (Active Comparator): MCT oil (20 g) was included in the test breakfast
  Interventions: Dietary Supplement: Test breakfast
- LCT (Placebo Comparator): Corn oil (20 g) was included in the test breakfast
  Interventions: Dietary Supplement: Test breakfast

INTERVENTIONS:
Dietary Supplement: Test breakfast

SUMMARY:
The purpose of this study is to test the effects of medium chain triglyceride consumption, relative to long chain triglycerides, on hormones involved in appetite regulation and food intake in overweight men. We expect medium chain triglycerides to reduce appetite and food intake and to do so by increasing levels of hormones known to be involved in satiety and reduce levels of those involved in appetite.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Weight stable (<10 lb over previous 3 months)
* Overweight (body mass index 25-29.9)

Exclusion Criteria:

* Smokers
* Excessive caffeine users
* Severe health conditions
* Allergy to food products/ingredients in the study
* Taking medications known to affect energy expenditure or gastrointestinal function

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Food intake | up to 3 hours
  Intake at an ad libitum meal 3 h after test oil consumption (Study 1) or 1 h after a pre-load containing the test oil (Study 2)

SECONDARY OUTCOMES:
Ghrelin | 3 hours
Peptide YY | 3 hours
Glucagon-like peptide 1 | 3 hours
Insulin | 3 hours
Triglycerides | 3 hours
Leptin | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — New York Obesity Nutrition Research Center
Locations (1):
- New York Obesity Nutrition Research Center, New York, New York, United States

REFERENCES:
- [Derived] St-Onge MP, Mayrsohn B, O'Keeffe M, Kissileff HR, Choudhury AR, Laferrere B. Impact of medium and long chain triglycerides consumption on appetite and food intake in overweight men. Eur J Clin Nutr. 2014 Oct;68(10):1134-40. doi: 10.1038/ejcn.2014.145. Epub 2014 Jul 30. PMID 25074387